

## **Statistical Analysis Plan**

### **VICTOR**

 $\underline{\textbf{\textit{V}}} \textbf{al}\underline{\textbf{\textit{I}}} \textbf{dation of } \underline{\textbf{\textit{C}}} \textbf{ardioMEMS HF Sys}\underline{\textbf{\textit{T}}} \textbf{em Cardiac} \underline{\textbf{\textit{O}}} \textbf{utput Algo}\underline{\textbf{\textit{R}}} \textbf{ithm IDE}$ 

NCT05428384

# Statistical Analysis Plan (SAP)

Version B

June 8, 2022



# Statistical Analysis Plan

### **TABLE OF CONTENTS**

| 1.0 | SYNOPSIS OF STUDY DESIGN | 4 |
|----------|------------------------------------------------------|----|
| 1.1 | Purpose of the Statistical Analysis Plan | 4 |
| 1.2 | Clinical Investigation Objectives | 4 |
| 1.3 | Clinical Investigation Design | 4 |
| 1.4 | Endpoints | 6 |
| 1.4 | 4.1 Primary Endpoint and Rationale | 6 |
| 1.4 | 4.2 Descriptive Endpoints | 6 |
| 1.5 | Blinding | 6 |
| 2.0 | ANALYSIS CONSIDERATIONS | 7 |
| 2.1 | Analysis Populations | 7 |
| 2. | 1.1 Enrolled Population | 7 |
| 2. | 1.2 Per Protocol (PP) Population | 7 |
| 2.2 | Statistical Methods | 7 |
| 2.2 | 2.1 Descriptive Statistics for Continuous Variables | 7 |
| 2.2 | 2.2 Descriptive Statistics for Categorical Variables | 7 |
| 2.3 | Endpoint Analysis | 7 |
| 2.3 | 3.1 Primary Endpoint | 7 |
| 2.4 | Sample Size Calculations | 8 |
| 2.5 | Interim Analysis | 9 |
| 2.6 | Timing of Analysis | 9 |
| 2.7 | Trial Success | 9 |
| 2.8 | Subgroups for Analysis | 9 |
| 2.9 | Handling of Missing Data | 9 |
| 2.10 | ) Poolability | 9 |
| 2.11 | Multiplicity | 9 |
| 2.12 | 2 Adjustments for Covariates | 10 |
| 3.0 | DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA | 10 |
| 3.1 | Baseline and Demographic Characteristics | 10 |
| 3.2 | Adverse Events | 10 |
| 3.3 | Subject Early Termination | 10 |
| 3.4 | Protocol Deviation | 10 |
| 3.5 | Descriptive Endpoints or Additional Data | 10 |
| 4.0 | DOCUMENTATION AND OHER CONSIDERATIONS | 12 |
| 5.0 | ACRONYMS AND ABBREVIATIONS | 12 |
| 379 Ver. | : G | |



| 6.0 | REFERENCES | 13 |
|-----|------------|----|
| 7.0 | APPENDICES | 14 |



### Statistical Analysis Plan

#### 1.0 SYNOPSIS OF STUDY DESIGN

#### 1.1 Purpose of the Statistical Analysis Plan

This statistical analysis plan (SAP) is intended to provide a detailed and comprehensive description of the planned methodology and analysis to be used for Clinical Investigational Plan (CIP) the Validation of CardioMEMS HF System Cardiac Output Algorithm (VICTOR) IDE clinical investigation. This plan is based on Version B Clinical Investigation Plan.

### 1.2 Clinical Investigation Objectives

There are two primary objectives of this clinical investigation. The first objective is to finalize development of the algorithm estimating CO by collecting paired cardiac Magnetic Resonance Imaging (cMRI) measurements of CO, as well as other parameters of heart function, and CardioMEMS HF System readings in the same subject. The second objective of this clinical investigation is to use data collected during the validation phase, distinct from the subjects within the development phase, to evaluate the agreement between the CardioMEMS HF System-derived CO and the CO values from cMRI CO values in patients previously implanted with the commercially available CardioMEMS HF System.

#### 1.3 Clinical Investigation Design





## Statistical Analysis Plan

Figure 1: Clinical Investigation Design



During validation, measurement data from a distinct subject cohort to subjects included in the development phase will be used to determine if the chosen algorithm meets the validation criteria.



designed this clinical investigation to involve as little pain, discomfort, fear, and any other foreseeable risk as possible for subjects. Refer to the Risk Analysis in Section 15.0 of this clinical investigation plan for details.



## Statistical Analysis Plan

#### 1.4 Endpoints

#### 1.4.1 Primary Endpoint and Rationale

The primary endpoint of this clinical investigation is to estimate CO from CardioMEMS HF System data. The estimated CO will be evaluated for agreement between the CardioMEMS HF System-derived CO and the CO values from cMRI in patients with the CardioMEMS HF System. Specifically, the primary endpoint will compare the two paired measurements taken at rest, collected during the 3-month follow-up visit from subjects allocated to the validation phase. Paired measurements will be compared using Deming regression. Agreement will be assessed through estimating the regression parameters of slope and intercept and evaluating their proximities to unity (slope=1 and intercept=0).



#### 1.4.2 Descriptive Endpoints

Paired measurements will be evaluated for the following data samples:

- Baseline measurements recorded at rest
- Baseline measurements recorded following introduction of Dobutamine
- 3) All Baseline measurements
- 4) 3 Month measurements recorded at rest
- 5) 3 Month measurements recorded following introduction of Dobutamine
- All 3 Month measurements
- 7) Baseline and 3 Month measurements recorded at rest
- 8) Baseline and 3 Month measurements recorded following introduction of Dobutamine
- 9) All Baseline and 3 Month measurements

Each data sample will be analyzed using Deming regression methods described for the primary endpoint, Bland-Altman methods, and relative error will be computed using the method proposed by Shoemaker et al.<sup>4</sup>

#### 1.5 Blinding

Investigators and subjects will not be blinded.



## Statistical Analysis Plan

#### 2.0 ANALYSIS CONSIDERATIONS

### 2.1 Analysis Populations

#### 2.1.1 Enrolled Population

The Enrolled population includes all enrolled subjects (development phase and validation phase),

- Informed Consent obtained
- Inclusion/Exclusion criteria satisfied

#### 2.1.2 Per Protocol (PP) Population



#### 2.2 Statistical Methods

#### 2.2.1 Descriptive Statistics for Continuous Variables

Continuous variables will be summarized with the numbers of observations, means and standard deviations, with quartiles, minimum and maximum.

#### 2.2.2 Descriptive Statistics for Categorical Variables

Categorical variables will be summarized with subject counts and percentages/rates.

#### 2.3 Endpoint Analysis

#### 2.3.1 Primary Endpoint

The primary endpoint of this clinical investigation is to estimate CO from CardioMEMS HF System data. The estimated CO will be evaluated for agreement between the CardioMEMS-derived CO and the CO values from cMRI in patients with the CardioMEMS HF System. Specifically, the primary endpoint will compare the two paired measurements taken at rest, collected during the 3-month follow-up visit from subjects allocated to the validation phase.



86379 Ver. G Template



## Statistical Analysis Plan



86379 Ver. G Template



### Statistical Analysis Plan



### 2.5 Interim Analysis

No formal interim analyses are planned for this study. As such, no formal statistical rule for early termination of the trial is defined.

## 2.6 Timing of Analysis

#### 2.7 Trial Success

The trial will be considered successful if Deming regression 95% confidence interval of the slope contains 1 and the 95% confidence interval of the intercept contains 0 for the primary endpoint.

#### 2.8 Subgroups for Analysis

There are no planned subgroup analyses for this trial.

### 2.9 Handling of Missing Data

The purpose of this trial is to validate an algorithm by comparing measurements using two methods. In order to evaluate the primary endpoint, a physical measurement must be recorded from each method, and thus, there is no planned sensitivity analysis or imputation procedure for missing data.

#### 2.10 Poolability

This trial is designed to be conducted in up to 15 centers in the United States. Given the sample size allocated for the primary endpoint, individual centers may not have adequate sample to assess individual center effect. Therefore, no formal poolability analysis is planned with overall results deemed poolable for interpretation of the study endpoints.

### 2.11 Multiplicity

This study includes a single primary endpoint. Thus, no Type I error adjustment is necessary.



## Statistical Analysis Plan

#### 2.12 Adjustments for Covariates

Unless otherwise specified, no adjustments for covariates will be made for any of the variables in the analyses.

### 3.0 <u>DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA</u>

### 3.1 Baseline and Demographic Characteristics

The following baseline and demographic variables will be summarized for the subjects in the Enrolled population: gender, age, ethnicity, race, cardiac disease history, medical history and co-morbidities, vital signs, and laboratory assessments.

#### 3.2 Adverse Events

Adverse events are defined in Section 7.1 of the Clinical Investigational Plan. All adverse events will be summarized for all subjects in the Enrolled population as number and percentage of all subjects who experience the event and the total number of events.

#### 3.3 Subject Early Termination

Subject early termination reasons including deaths, withdrawals, lost-to-follow-up, etc. will be summarized by analysis population at all scheduled visits.

#### 3.4 Protocol Deviation

Protocol deviations will be summarized by major and minor categories for subjects in whom a protocol deviation was reported.

#### 3.5 Descriptive Endpoints or Additional Data

Descriptive endpoints will evaluate data for the following data samples:

- 1) Baseline measurements recorded at rest
- 2) Baseline measurements recorded following introduction of Dobutamine
- 3) All Baseline measurements
- 4) 3 Month measurements recorded at rest
- 5) 3 Month measurements recorded following introduction of Dobutamine
- 6) All 3 Month measurements
- 7) Baseline and 3 Month measurements recorded at rest
- 8) Baseline and 3 Month measurements recorded following introduction of Dobutamine
- 9) All Baseline and 3 Month measurements







## Statistical Analysis Plan

### 4.0 **DOCUMENTATION AND OHER CONSIDERATIONS**

## 5.0 ACRONYMS AND ABBREVIATIONS

| Acronym or Abbreviation | Complete Phrase or Definition |
|-------------------------|------------------------------------|
| CI | Confidence Interval |
| cMRI | Cardiac Magnetic Resonance Imaging |
| CIP | Clinical Investigation Plan |
| CO | Cardiac Output |
| MRI | Magnetic Resonance Imaging |
| OLR | Ordinary Least-squares Regression |
| SAP | Statically Analysis Plan |
| SDa | Analytical Standard Deviation |



## Statistical Analysis Plan

#### 6.0 **REFERENCES**

- Critchley, L.A.H., Critchley, J.A.J.H. A Meta-Analysis of Studies Using Bias and Precision Statistics to Compare Cardiac Output Measurement Techniques. J Clin Monit Comput 15, 85–91 (1999). https://doi.org/10.1023/A:1009982611386
- 2. Linnet K. Necessary sample size for method comparison studies based on regression analysis. Clin Chem. 1999 Jun;45(6 Pt 1):882-94. PMID: 10351998.
- 3. Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID: 10501650.
- Shoemaker WC, Wo CC, Bishop MH, Appel PL, Van de Water JM, Harrington GR, Wang X, Patil RS. Multicenter trial of a new thoracic electrical bioimpedance device for cardiac output estimation. Crit Care Med. 1994 Dec;22(12):1907-12. PMID: 7988125.
- 5. Deal, AM, Pate, VW, Rouby, SE, A SAS Macro for Deming Regression, Presented at Southeast SAS Users Group (SESUG) 2009, http://analytics.ncsu.edu/sesug/2009/CC014.Deal.pdf.
- 6. Tree, M., White, J., Midha, P., Kiblinger, S., and Yoganathan, A. (November 5, 2015). "Validation of Cardiac Output as Reported by a Permanently Implanted Wireless Sensor." ASME. J. Med. Devices. March 2016; 10(1): 011001. https://doi.org/10.1115/1.4031799
- 7. Hoeper MM, Maier R, Tongers J, Niedermeyer J, Hohlfeld JM, Hamm M, Fabel H. Determination of cardiac output by the Fick method, thermodilution, and acetylene rebreathing in pulmonary hypertension. Am J Respir Crit Care Med. 1999 Aug;160(2):535-41. doi: 10.1164/ajrccm.160.2.9811062. PMID: 10430725.
- Dhingra VK, Fenwick JC, Walley KR, Chittock DR, Ronco JJ. Lack of agreement between thermodilution and fick cardiac output in critically ill patients. Chest. 2002 Sep;122(3):990-7. doi: 10.1378/chest.122.3.990. PMID: 12226045.
- 9. Gonzalez J, Delafosse C, Fartoukh M, Capderou A, Straus C, Zelter M, Derenne JP, Similowski T. Comparison of bedside measurement of cardiac output with the thermodilution method and the Fick method in mechanically ventilated patients. Crit Care. 2003 Apr;7(2):171-8. doi: 10.1186/cc1848. Epub 2002 Dec 20. PMID: 12720564; PMCID: PMC270608.
- Baylor P. Lack of agreement between thermodilution and fick methods in the measurement of cardiac output. J Intensive Care Med. 2006 Mar-Apr;21(2):93-8. doi: 10.1177/0885066605285234. PMID: 16537751.
- Weinbroum AA, Biderman P, Soffer D, Klausner JM, Szold O. Reliability of cardiac output calculation by the fick principle and central venous oxygen saturation in emergency conditions. J Clin Monit Comput. 2008 Oct;22(5):361-6. doi: 10.1007/s10877-008-9143-y. Epub 2008 Oct 23. PMID: 18946716.
- Fares WH, Blanchard SK, Stouffer GA, Chang PP, Rosamond WD, Ford HJ, Aris RM. Thermodilution and Fick cardiac outputs differ: impact on pulmonary hypertension evaluation. Can Respir J. 2012 Jul-Aug;19(4):261-6. doi: 10.1155/2012/261793. PMID: 22891186; PMCID: PMC3411391.
- 13. Rich JD, Archer SL, Rich S. Noninvasive cardiac output measurements in patients with pulmonary hypertension. Eur Respir J. 2013 Jul;42(1):125-33. doi: 10.1183/09031936.00102212. Epub 2012 Oct 25. PMID: 23100501.
- Bland, J & Altman, Douglas. (2007). Agreement Between Methods of Measurement with Multiple Observations Per Individual. Journal of biopharmaceutical statistics. 17. 571-82. 10.1080/10543400701329422.



# Statistical Analysis Plan

## 7.0 APPENDICES





## Statistical Analysis Plan

### **APPENDIX B: SAMPLE SIZE CALCULATION DETAILS**



86379 Ver. G Template























# Statistical Analysis Plan

### APPENDIX D: STATISTICAL ANALYSIS PLAN REVISIONS



86379 Ver. G Template



| Ver | Details | Rationale |
|-----|---------|-----------|